CLINICAL TRIAL: NCT05578274
Title: Abscopal Effect from the Addition of Low-dose Radiotherapy in Metastatic Cancer Patients Receiving Stereotactic Body Radiotherapy: a Multicenter, Randomized Clinical Study
Brief Title: Abscopal Effect from Low-dose Radiotherapy in Metastatic Cancer Combined with Stereotactic Body Radiotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Ah Ram Chang, Director of Radiation Oncology, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHUH 2022-07-004-001
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms; Secondary Malignant Neoplasm
Keywords: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBRT+LDRT (Experimental): In the experimental group, stereotactic body radiotherapy (SBRT) and low-dose radiotherapy (LDRT) are administered concurrently. SBRT is administered three times, at intervals of 1-2 days, with LDRT. LDRT is planned to irradiate EQD2 6 Gy considering the scattered dose caused by SBRT.
  Interventions: Radiation: SBRT + LDRT
- SBRT alone (Active Comparator): In the control group, stereotactic body radiotherapy (SBRT) alone is performed. SBRT is administered three times, at intervals of 1-2 days. The scattered dose should not exceed EQD2 2Gy to the non-irradiated lesion.
  Interventions: Radiation: SBRT alone

INTERVENTIONS:
Radiation: SBRT + LDRT — SBRT is performed according to the protocol of each institution. However, the total fraction of SBRT is fixed to 3, and the treatment interval is maintained for 1-2 days.
  The scattered dose should not exceed EQD2 (α/β=10) 2 Gy for non-irradiated lesions.
  LDRT is planned to irradiate EQD2 (α/β=10) 6 Gy to lesions, considering the scattered dose caused by SBRT.
  If there are non-irradiated lesions, they are defined as internal control, and the total dose is limited to 0.5 Gy or less.
  CTV allows up to 5 mm margin for GTV, and 3-10mm for PTV margin from CTV. It is planned that the iso-dose line corresponding to the prescribed dose contains at least 90% of PTV and 95% of GTV.
  Arms: SBRT+LDRT
Radiation: SBRT alone — SBRT is performed according to the protocol of each institution. However, the total fraction of SBRT is fixed to 3, and the treatment interval is maintained for 1-2 days.
  The scattered dose should not exceed EQD2 (α/β=10) 2 Gy for non-irradiated lesions.
  Arms: SBRT alone

SUMMARY:
Stereotactic body radiotherapy (SBRT) has been known to enhance the abscopal effect by up to 40% when delivered with immune checkpoint inhibitors (ICIs). Recently, preclinical and clinical studies demonstrate that metastatic lesions treated with non-cytotoxic low-dose radiotherapy (LDRT) significantly were reduced in the condition where SBRT and ICIs were administered together. Given that ICIs are highly expensive and some tumors are beyond the indications of ICIs, novel approaches are required to boost the abscopal effect in the absence of ICIs. Therefore, the investigators design a multicenter, randomized clinical trial that investigates the efficacy and safety of LDRT combined with SBRT in metastatic cancer patients. The primary endpoint is a lesion-specific response of LDRT lesions (i.e., abscopal effect) evaluated three months after radiotherapy.

Subjects will be randomly allocated into two groups (1:1) with the stratification by planning target volume and previous use of ICIs: control group (SBRT in three fractions) or experimental group (SBRT + LDRT in three factions). Unless patients agree with randomization, subjects will participate in a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Randomization study: Patients who can provide their written informed consent
* Cohort study: Patients who do not consent to randomization and who are able to consent to a prospective cohort study and provide written informed consent
* Age ≥19 years
* Patients with histologically confirmed primary solid (irrespective of the status of the primary tumor)
* Patients with ECOG performance status 0-2
* Patients planning stereotactic body radiotherapy for extracranial metastases
* Based on RECIST v1.1, patients with at least one extracranial measurable lesion other than SBRT lesions
* Patients with one or more measurable lesions, which are not suitable for SBRT or palliative radiotherapy and can be considered for LDRT (bone metastasis is not indicated for LDRT)
* Patients with hematologic function suitable for radiotherapy (absolute neutrophil count ≥1,500/mm^3, hemoglobin ≥9 g/dL, platelet count ≥100,000/mm^3)
* Patients with a life expectancy of 6 months or more according to the researcher's judgment

Exclusion Criteria:

* Patients participating in other clinical studies that may affect the efficacy/safety of this clinical study
* Patients with brain metastasis
* Patients planning SBRT for all measurable lesions due to oligometastasis
* Patients with a history of radiotherapy for extracranial metastases within 3 months of the enrollment
* Patients unable to cooperate with stereotactic body radiotherapy
* Patients who are pregnant or planning to
* Patients with advanced or multiple malignancies requiring aggressive treatment (excluding skin cancers other than melanoma or intraepithelial cancer)
* Patients who have received systemic steroid therapy or immunosuppressive therapy within 2 weeks of enrollment - Patients with an (e.g. allergic disease, radiation pneumonitis, etc.) active autoimmune disease requiring systemic treatment within the past 2 years, evidence of clinically severe autoimmune disease, or syndrome requiring systemic steroid or immunosuppressive therapy (Patients who need intermittent use of bronchodilators, inhaled steroids, or topical steroid injections, hypothyroid patients on stable hormone replacement therapy, type 1 diabetes patients, or patients recovering from childhood asthma/atopic dermatitis are permitted)
* Patients with active infection requiring systemic treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Abscopal effect rate of low-dose radiotherapy lesions | 3 months after completion of radiotherapy

SECONDARY OUTCOMES:
Abscopal effect rate of low-dose radiotherapy lesions | 1, 6, and 12 months after completion of radiotherapy
Overall response rate | 1, 3, 6, and 12 months after completion of radiotherapy

OTHER OUTCOMES:
Progression-free survival rate | 12 months after completion of radiotherapy
Overall survival rate | 12 months after completion of radiotherapy
Adverse event | up to 12 months after completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ah Ram Chang, MD, PhD, Study Chair — Soonchunhayng Universtiy Seoul Hospital